CLINICAL TRIAL: NCT02088268
Title: Treatment and Evaluation of Platelet-rich-plasma on Diabetes Wound Healing
Brief Title: Treatment of PRP on Diabetes Wound
Acronym: PRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH102-REC1-110
Record Dates: First submitted 2014-01-21; First posted 2014-03-14 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Diabetic Ulcers on Both Feet
MeSH Terms: interventions — Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- platelet-rich plasma (Experimental): wound healing
  Interventions: Other: wound healing

INTERVENTIONS:
Other: wound healing — wound healing

SUMMARY:
The purpose of this study is to focus on the effect of platelet-rich-plasma on diabtic ulcer foot, as adjuvant treatment along with the standard care of chronic diabetic, and evaluate the efficiency and the clinical application of PRP on serious wound healing.

DETAILED DESCRIPTION:
Diabetes is a condition in which the body dose not effectively use sugar so that there is too much sugar in the blood. It is estimated that 15% of the diabetics suffer from diabetic food ulcers at some point. The healing process can be slow and easily to be infected with some pathogens so the patients are at risk in amputation. The wound healing process is a complex mechanism involves the interaction of molecular signals and different cell types. Platelets play important roles in wound healing. When injury occurs platelets are activated with thrombin and clot is formed. In addition to the function of hemostasis, activated platelets release many growth factors that trigger angiogenesis, extracellular matrix production and cytokine release, which is need for wound healing.

Platelet-rich plasma (PRP) is a portion of plasma fraction of autologous blood having a high concentration of thrombocytes. Thrombin induces the activation of PRP and results in the release of multiple growth factors, including platelet-derived growth factor (PDGF), vascular endothelial growth factor (VEGF), epidermal growth factor (EGF), insulin-like growth factor (IGF), and transforming growth factor beta (TGF-β). PRP is known for the capacity to stimulate cell proliferation and differentiation. PRP can also interact with macrophage to improve tissue healing and regeneration, and exhibit potent activities against several kinds of pathogens.

Our study will focus on the advantage of PRP for aiding wound healing for diabetes. PRP from autologous blood can be mixed with thrombin in appropriate ratio and inject into the sites around the wound, as adjuvant treatment along with the standard care of chronic diabetic. The wound will be checked 1 to 2 times each week for the evaluation of PRP on clinical application.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patient who suffers from sereious alcer feet.
* age of 20-70 years old

Exclusion Criteria:

* patient with systemic disorder
* psycho
* patient with coagulation abnormality
* patient with inflammation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
effect of PRP on diabete wound closure | every 2 weeks, from the first date of PRP treatment and up to 12 weeks.
  The wound was checked twicw each month using a digital camera and ruler to trace the area of wound. Wound closure was determined as the percentage closed and calculated as:
  % Closed = [（Area on Day 0 - Open Area on Final Day）] x 100

CONTACTS AND LOCATIONS:
Overall Officials: Jeng Long-Bin, Study Chair — organ transplantation center
Locations (1):
- China Medical University Hospital, Taichung, Taiwan